CLINICAL TRIAL: NCT02629354
Title: A Single Center, Single Dose, Open Label, Randomized, Two Period, Two Sequence Crossover Study to Evaluate the Relative Bioavailibility of Ibuprofen From a Fixed-dose Combination Tablet Containing Ibuprofen 400 mg and Caffeine 100 mg and a Tablet of Ibuprofen 400 mg in at Least 30 Healthy Males and Females Under Fed Conditions
Brief Title: To Determine Blood Concentrations of Ibuprofen and Caffeine in a Tablet Against Ibuprofen Alone From Another Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1335.3
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — Ibuprofen; Caffeine

ARMS (2):
- Ibuprofen and Caffeine (Experimental)
  Interventions: Drug: Ibuprofen; Drug: Caffeine
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen
  Arms: Ibuprofen and Caffeine
Drug: Caffeine
  Arms: Ibuprofen and Caffeine
Drug: Ibuprofen
  Arms: Ibuprofen

SUMMARY:
The objective of the trial is to compare to combination of 400 mg ibuprofen and 100 mg caffeine against 400 mg ibuprofen alone under fed conditions

ELIGIBILITY:
Inclusion criteria:

* Healthy males and females, 18 to 50 years (inclusive) at time of screening.
* Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 (inclusive).
* Body mass not less than 50 kg.
* Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the PI considers the deviation to be irrelevant for the purpose of the study.
* Non-smokers and mild or moderate smokers (<= 10 cigarettes or pipes per day). Further inclusion criteria apply

Exclusion criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females. One unit is equal to beer [200 mL/10 ounces], wine [100 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Regular exposure to substances of abuse (other than alcohol) within the past year.
* Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks before the first administration of IMP except if this will not affect the outcome of the study in the opinion of the PI. In this study the concomitant use of hormonal contraceptives is allowed.
* Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks (or within 5 elimination half-lives for chemical entities or 2 elimination half-lives for anti-bodies or insulin), whichever is the longer) before administration of IMP in this study, at the discretion of the PI.
* Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
* History of hypersensitivity or allergy (angioedema or urticaria) to the IMP or its excipients or any related medication (Aspirin or any other NSAID).
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
* Renal impairment.
* Positive urine screen for drugs of abuse. In case of a positive result the urine screen for drugs of abuse may be repeated once at the discretion of the PI.

Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Bloemfontein, South Africa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended a specialist site ensured that they (the subjects) met all inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- Ref - Test: Subjects received the reference product (Ref) which was a single oral dose (1 film-coated tablet) of 400 milligram (mg) ibuprofen (equivalent to 684 mg ibuprofen lysinate, trade name: Dolormin® Extra) under fed conditions. After a washout period of at least 6 calendar days, the subjects received the test product (Test), which was a single oral dose of 400 mg ibuprofen acid and 100 mg caffeine in a film coated tablet as a fixed dose combination (FDC), under fed conditions. Finally the subjects had a follow-up phase of 72 hours.
- Test - Ref: Subjects received the test product (Test) which was a single oral dose of 400 mg ibuprofen acid and 100 mg caffeine in a film coated tablet as a FDC under fed conditions. After a washout period of at least 6 calendar days, the subjects received the reference product (Ref), which was a single oral dose (1 film-coated tablet) of 400 milligram (mg) ibuprofen (equivalent to 684 mg ibuprofen lysinate, trade name: Dolormin® Extra), under fed conditions. Finally the subjects had a follow-up phase of 72 hours.
Period: Period 1
Arm/Group | Ref - Test | Test - Ref
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Ref - Test | Test - Ref
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Ref - Test | Test - Ref
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Ref - Test | Test - Ref
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population: all subjects randomized to a treatment sequence.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ref - Test | Test - Ref | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (8.49) | 26.1 (5.59) | 28.0 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of S-ibuprofen
Description: This outcome measure presents the maximum observed concentration (Cmax) of S-ibuprofen in plasma obtained directly from the concentration-time data.
Time Frame: Within 2 hours prior to dosing and at 5, 10,15, 30 and 45 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose
Population: Pharmacokinetic (PK) population: all subjects who completed the PK sampling in both periods and with no major protocol deviations considered to impact on the analysis of the PK data were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/ millilitre (mL)
Groups:
- Reference Product: Subjects received a single oral dose of 400 mg ibuprofen (trade name: Dolormin® Extra), under fed condition.
- Test Product: Subjects received a single oral dose of 400 mg ibuprofen acid and 100 mg caffeine as a FDC under fed condition.
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 26 | 26
nanogram (ng)/ millilitre (mL) | 13268.7 (38.0) | 14967.2 (34.9)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; Relative bioavailability [%] was estimated by the ratios of the geometric means (100*test/reference [T/R]). Additionally, it's two-sided 90% confidence interval (CI) was provided; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 113.77, 90% CI 2-sided [98.99 to 130.75] — Analysis of variance (ANOVA) with fixed effects for sequence, subject nested within sequence, period and product after logarithmic transformation of the data

2. Primary Outcome: Cmax of R-ibuprofen
Description: This outcome measure presents the Cmax of R-ibuprofen in plasma obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 26 | 26
ng/mL | 10495.7 (32.7) | 11454.6 (26.6)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; Relative bioavailability [%] was estimated by the ratios of the geometric means (100*test/reference [T/R]). Additionally, it's two-sided 90% CI was provided; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 110.16, 90% CI 2-sided [96.32 to 125.97] — ANOVA with fixed effects for sequence, subject nested within sequence, period and product after logarithmic transformation of the data

3. Primary Outcome: Cmax of Ibuprofen
Description: This outcome measure presents the Cmax of ibuprofen in plasma obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 26 | 26
ng/mL | 23557.9 (34.8) | 26309.5 (30.3)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 112.69, 90% CI 2-sided [98.49 to 128.94] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Area Under the Plasma Concentration of S-ibuprofen Versus Time Curve, From Time Zero to t (AUC0-t)
Description: This outcome measure presents the area under the plasma concentration of S-ibuprofen versus time curve, from time zero to t, where t is the time of the last quantifiable concentration (AUC0-t).
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)*ng/mL
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 26 | 26
hour (h)*ng/mL | 65110 (21.9) | 63150 (21.7)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 97.36, 90% CI 2-sided [94.61 to 100.19] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Area Under the Plasma Concentration of S-ibuprofen Versus Time Curve, With Extrapolation to Infinity (AUC0-INF)
Description: This outcome measure presents the area under the plasma concentration of S-ibuprofen versus time curve, with extrapolation to infinity (AUC0-INF).
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 25 | 26
h*ng/mL | 68900 (17.2) | 64990 (20.6)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 96.47, 90% CI 2-sided [93.74 to 99.28] — [estimate comment as in outcome 2, analysis 1]

6. Primary Outcome: AUC0-t of R-ibuprofen
Description: This outcome measure presents the area under the plasma concentration of R-ibuprofen versus time curve, from time zero to t, where t is the time of the last quantifiable concentration (AUC0-t).
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 26 | 26
h*ng/mL | 42480 (19.0) | 41200 (15.9)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 97.55, 90% CI 2-sided [92.57 to 102.80] — [estimate comment as in outcome 2, analysis 1]

7. Primary Outcome: AUC0-t of Ibuprofen
Description: This outcome measure presents the area under the plasma concentration of ibuprofen versus time curve, from time zero to t, where t is the time of the last quantifiable concentration (AUC0-t).
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 26 | 26
h*ng/mL | 108400 (18.4) | 105300 (16.9)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 97.57, 90% CI 2-sided [94.50 to 100.73] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: AUC0-INF of R-ibuprofen
Description: This outcome measure presents the area under the plasma concentration of R-ibuprofen versus time curve, with extrapolation to infinity (AUC0-INF).
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 25 | 26
h*ng/mL | 43910 (17.2) | 41960 (16.3)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 97.21, 90% CI 2-sided [92.22 to 102.46] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: AUC0-INF of Ibuprofen
Description: This outcome measure presents the area under the plasma concentration of ibuprofen versus time curve, with extrapolation to infinity (AUC0-INF).
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product | Test Product
Number analyzed (Participants) | 25 | 26
h*ng/mL | 113200 (14.6) | 107300 (16.4)
Statistical Analysis 1: Comparison: Reference Product vs Test Product; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Percent Ratio Test/Ref = 96.83, 90% CI 2-sided [93.75 to 100.01] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From first administration of study medication until 3 days after last dosing (up to 11 days).
Arm/Group | Reference Product | Test Product
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.